CLINICAL TRIAL: NCT01054612
Title: Tissue Sectioning by Electro-Dissociation
Status: Withdrawn | Type: Observational
Why Stopped: The study was closed due to the departure of several of the co-investigators.
Sponsor: University of Arkansas (Other)
Responsible Party: Dr. Gal Shafirstein, University of Arkansas, Arkansas Children's Hospital
Other Study IDs: IRB 28177; NBIB
Record Dates: First submitted 2007-12-21; First posted 2010-01-22 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Thin Sections; Fresh Unfixed Tissues; Fresh Unfrozen Tissues
Keywords: Histology; Immunohistochemical; Gene Expression; Tissue Sectioning

INTERVENTIONS:
Other: Tissue Sectioning via Electro Erosion Process — Focused RF energy can be used to produce consecutive thin sections of fresh tissue for immunohistochemical and nucleic acids analysis by electro-dissociation without thermal damage, ultimately allowing high resolution reconstruction of gene and protein expression patterns of large tissue specimens in 3D.

SUMMARY:
Currently there is no technique to produce thin (0.004-0.01 mm) serial sections of large fresh tissue specimens that are suitable for high-resolution in situ protein/gene expression studies without ice artifact or fixation-induced molecular damage. Traditional frozen sectioning preserves protein and nucleic acid structure, but the inherent ice artifact precludes reconstruction of protein and mRNA expression patterns in 3-dimensions. Since the limitations of the existing sectioning techniques result from the fact that they rely on mechanical cutting which in turn require the tissue to be stiff, we suggest a new approach to cut tissue via an electro erosion process that utilizes focus radio frequency (RF).

ELIGIBILITY:
Inclusion Criteria:

* Fresh Tissue
* Unfrozen Tissue
* Unfixed Tissue

Exclusion Criteria:

* Unfresh Tissue
* Frozen Tissue
* Fixed Tissue

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Discarded human tissue obtained immediately following surgical resection
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gal Shafirstein, Ph.D., Principal Investigator — UAMS, ACH, Central Arkansas Veterans Healthcare System